CLINICAL TRIAL: NCT02821871
Title: the Food Effect Pharmacokinetic, Material Balance and Metabolite Identification of SP2086 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SP2086-110
Record Dates: First submitted 2016-06-26; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, High-Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SP2086 (Active Comparator): All subjects were ransomed to A and B sequence.In A sequence,subjects take SP2086 100mg once in fasting the first day,and the B sequence subjects need to take SP2086 100mg after the high fat diet.In Day 8，the medicine strategy of two sequence subjects were alternately.
  Interventions: Dietary Supplement: high fat diet
- high fat diet (Other): All subjects were ransomed to A and B sequence.In A sequence,subjects take SP2086 100mg once in fasting the first day,and the B sequence subjects need to take SP2086 100mg after the high fat diet.In Day 8，the medicine strategy of two sequence subjects were alternately.
  Interventions: Drug: SP2086

INTERVENTIONS:
Drug: SP2086
  Arms: high fat diet
Dietary Supplement: high fat diet
  Arms: SP2086

SUMMARY:
All eligible subjects were randomly assigned to group A and group B sequences, each sequence has 12 subjects. The SP2086 were given limosis,then after the meal,then limosis.In the study ,the investigators collected the blood samples,urine samples and fecal samples to analyze.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index (BMI, a measure of a person's weight in relation to height) between 19 and 26 kg/m2

Exclusion Criteria:

* History of diabetes
* History of heart failure or renal insufficiency
* Urinary tract infections, or vulvovaginal mycotic infections
* History of or current clinically significant medical illness as determined by the Investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose
* Known allergy to SP2086 or any of the excipients of the formulation of SP2086

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SP2086 | up to Day 12
  Cmax (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of SP2086
The maximum plasma concentration (Cmax) of SP2086 acid | up to Day 12
  Cmax (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of a single dose of SP2086.
The area under the plasma concentration-time curve (AUC) of SP2086 | up to Day 12
  AUC (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of SP2086.
The area under the plasma concentration-time curve (AUC) of SP2086 acid | up to Day 12
  AUC (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of a single dose of SP2086.
Cumulative percentage drainage of SP2086 in urine | up to Day 12
Cumulative percentage drainage of SP2086 in fecal | up to Day 12

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China